CLINICAL TRIAL: NCT06133465
Title: Pure Florid and Pleomorphic Lobular Carcinoma in Situ of the Breast: Towards an Increasingly Uniform Management. A Multicenter Observational Retrospective Study.
Brief Title: Pure Florid and Pleomorphic Lobular Carcinoma in Situ of the Breast: Towards an Increasingly Uniform Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Ferrucci Massimo, Principal Investigator, MD PhD, Istituto Oncologico Veneto IRCCS
Other Study IDs: 22171
Record Dates: First submitted 2023-11-02; First posted 2023-11-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pleomorphic Lobular Breast Carcinoma in Situ; Breast Florid Lobular Carcinoma in Situ
MeSH Terms: interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pleomorphic Lobular Carcinoma in Situ (PLCIS) of the breast: Patients with diagnosis of pure pleomorphic lobular carcinoma in situ of the breast
  Interventions: Procedure: Surgical wide local excision; Procedure: Cavity shaving; Procedure: Excision margin surgical clearance; Radiation: Adjuvant Radiotherapy; Biological: Adjuvant Hormone Therapy
- Florid Lobular Carcinoma in Situ (FLCIS) of the breast: Patients with diagnosis of pure florid lobular carcinoma in situ of the breast
  Interventions: Procedure: Surgical wide local excision; Procedure: Cavity shaving; Procedure: Excision margin surgical clearance; Radiation: Adjuvant Radiotherapy; Biological: Adjuvant Hormone Therapy

INTERVENTIONS:
Procedure: Surgical wide local excision — Surgical excision of breast carcinoma
Procedure: Cavity shaving — Cavity shaving of resection margins to guarantee oncological safety
Procedure: Excision margin surgical clearance — Surgical clearance of involved and/or closed excision margins
Radiation: Adjuvant Radiotherapy — Adjuvant radiotherapy
Biological: Adjuvant Hormone Therapy — Adjuvant hormone therapy

SUMMARY:
The goal of this retrospective multicenter observational study is to understand and evaluate the diagnostic and therapeutic management of pure forms of Florid Lobular Carcinoma In Situ (FLCIS) and Pleomorphic Lobular Carcinoma In Situ (PLCIS) of the breast. It addresses the significant challenges and controversies surrounding their clinical management, due to a lack of consensus or approved international guidelines.

The main questions this study aims to answer are:

* How is the diagnostic process for pure FLCIS and PLCIS currently managed?
* What are the primary therapeutic approaches for these specific breast conditions?
* How are positive and "close" surgical excision margins handled?
* Is adjuvant treatment, such as hormone therapy and radiotherapy, necessary?
* What factors are associated with recurrences?
* What are the rates of recurrences and/or upgrade to invasive carcinoma?

Participants will retrospectively collect all cases of pure FLCIS and PLCIS, reporting detailed data about their diagnostic and therapeutic management, as well as clinical and survival outcomes.

Methodology:

This international multicenter retrospective study will collect cases involving the pure forms of FLCIS and PLCIS of the breast. The study aims to provide insights into the current diagnostic and therapeutic approaches, along with the identification of opportunities to enhance clinical management, ultimately providing evidence-based recommendations and addressing the current lack of scientific literature regarding their treatment.

DETAILED DESCRIPTION:
Classical lobular carcinoma in situ (CLCIS) of the breast is considered a non-obligate precursor of invasive carcinoma. Histologically, it is categorized as a lesion with uncertain malignancy potential, and clinical management often parallels that of benign neoplastic conditions.

In contrast, its two variants, florid LCIS (FLCIS) and pleomorphic LCIS (PLCIS), have distinct morphological and genetic characteristics and a higher probability of being obligatory precursors to invasive carcinoma.

PLCIS shows marked cellular-nuclear pleomorphism, resembling high-grade ductal carcinoma in situ (often initially misdiagnosed as such).

FLCIS, on the other hand, displays a complete architectural subversion of lobular structure due to the increased rate of cell replication.

Both variants may show foci of comedonecrosis, a distinctive but not specific diagnostic feature.

A significant difference from CLCIS is their breast distribution; CLCIS tends to be multifocal, while the two variants typically present as unifocal.

Genetically, the two variants differ from CLCIS, with higher genetic instability, and increased alterations in genes coding for tumor suppressors and proteins involved in cell growth regulation and replication.

Immunohistochemically, both FLCIS and PLCIS regularly express estrogen and progesterone receptors, and they may present higher HER2 (Human Epidermal growth factor Receptor 2 - ERBB2 gene) over-expression compared to CLCIS.

Many controversies persist in the clinical management of these variants, largely due to their rarity in pure, isolated forms. Often, they are associated with an invasive carcinoma, which becomes the primary therapeutic focus, according to well established treatment protocols. Dedicated studies, both prospective and retrospective, are completely lacking in the literature, especially for pure FLCIS. Consequently, there is no consensus or approved international guidelines for accurate diagnostic-therapeutic strategies. Even the histological categorization of biopsy tests still remains a subject of debate.

Presently, there is unanimous consensus on the indication for surgical excision of these lesions to improve histological definition and exclude the presence of an invasive neoplastic focus. However, there is no consensus on the need of surgical margins cavity shaving and the management of resection margins when they are proved to be close or involved at the final specimen pathological report. Furthermore, there is a lack of evidence-based recommendations for adjuvant therapies like radiotherapy or endocrine therapy. Some scientific international associations, such as ESMO (European Society of Medical Oncology), suggest a similar approach to pleomorphic variants as for ductal carcinoma in situ due to their morphological similarity; yet, in the absence of robust evidence, this stance does not definitively support the benefit of adjuvant therapeutic strategies and poses a relative risk of overtreatment.

To address these challenges, the investigators propose international multicenter retrospective collection of cases involving the pure forms of FLCIS and PLCIS. Our goal is to comprehensively analyze the diagnostic and therapeutic management of this specific patient group and, notably, to fill the gap in the scientific literature regarding their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of PLCIS and/or FLCIS of the breast on both core-biopsy and/or on final specimen histology;
* Aged 18 years or older.

Exclusion Criteria:

* Histologic diagnosis of CLCIS;
* Histologic diagnosis of LCIS (any type) associated with invasive carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pure variant pleomorphic and/or florid lobular carcinoma in situ of the breast
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | From date of surgery until the date of first documented recurrence, assessed up to 120 months
  Recurrence rate (both invasive and LCIS, any type)
Upgrade rate to invasive carcinoma | From date of diagnostic core biopsy until the date of final pathology report after surgery, assessed up to 6 months
  Upgrade rate from PLCIS and/or FLCIS to invasive carcinoma from diagnostic core-biopsy to final specimen histology

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of surgery until the date of last follow-up or date of death from any cause, whichever came first, assessed up to 120 months
Disease-free survival (DFS) | From date of surgery until the date of first recurrence, whenever occurred, assessed up to 120 months
Rate of re-operation and/or radiotherapy boost and/or clinical follow-up after "close" or involved resection margins being reported | From date of surgery until the date of surgical margins management completion (any potential clinical follow-up included), assessed up to 72 months
  Management of involved and/or closed surgical resection margins
Postoperative complications | From date of surgery until any post-operative complications are resolved, assessed up to 3 months
  Incidence and management of post-operative complications
Rate of adjuvant therapies utilization | From date of surgery until the date of adjuvant therapies completion, assessed up to 120 months
  Adjuvant therapies and associated side effects

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Ferrucci, MD PhD, Principal Investigator — Istituto Oncologico Veneto IRCCS
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy

REFERENCES:
- [Background] Lakhani S, Schnitt S, O'Malley F, et al. Lobular neoplasia. In: Lakhani S, Ellis I, Schnitt S, Tan P, van de Vijer M, eds. WHO Classification of Tumours of the Breast, 2nd ed. Lyon, France: International Agency for Research on Cancer; 2012:77-80
- [Background] Page DL, Schuyler PA, Dupont WD, Jensen RA, Plummer WD Jr, Simpson JF. Atypical lobular hyperplasia as a unilateral predictor of breast cancer risk: a retrospective cohort study. Lancet. 2003 Jan 11;361(9352):125-9. doi: 10.1016/S0140-6736(03)12230-1. PMID 12531579
- [Background] Wen HY, Brogi E. Lobular Carcinoma In Situ. Surg Pathol Clin. 2018 Mar;11(1):123-145. doi: 10.1016/j.path.2017.09.009. Epub 2017 Dec 8. PMID 29413653
- [Background] Frost, A. R., T. N.Tsangaris, and S. G.Silverberg. Pleomorphic lobular carcinoma in situ. Pathol Case Rev 1996. 1:27-31.
- [Background] Sneige N, Wang J, Baker BA, Krishnamurthy S, Middleton LP. Clinical, histopathologic, and biologic features of pleomorphic lobular (ductal-lobular) carcinoma in situ of the breast: a report of 24 cases. Mod Pathol. 2002 Oct;15(10):1044-50. doi: 10.1097/01.MP.0000027624.08159.19. PMID 12379750
- [Background] Shin, S. J., R. A.DeLellis, D. M.Knowles, et al. "Florid" lobular carcinoma in situ with necrosis and calcification: a clinicopathologic, immunohistochemical and molecular analysis. Mod Pathol 2002. 15:52A.
- [Background] Shin SJ, Lal A, De Vries S, Suzuki J, Roy R, Hwang ES, Schnitt SJ, Waldman FM, Chen YY. Florid lobular carcinoma in situ: molecular profiling and comparison to classic lobular carcinoma in situ and pleomorphic lobular carcinoma in situ. Hum Pathol. 2013 Oct;44(10):1998-2009. doi: 10.1016/j.humpath.2013.04.004. Epub 2013 Jun 25. PMID 23809857
- [Background] Vos CB, Cleton-Jansen AM, Berx G, de Leeuw WJ, ter Haar NT, van Roy F, Cornelisse CJ, Peterse JL, van de Vijver MJ. E-cadherin inactivation in lobular carcinoma in situ of the breast: an early event in tumorigenesis. Br J Cancer. 1997;76(9):1131-3. doi: 10.1038/bjc.1997.523. PMID 9365159
- [Background] Bratthauer GL, Moinfar F, Stamatakos MD, Mezzetti TP, Shekitka KM, Man YG, Tavassoli FA. Combined E-cadherin and high molecular weight cytokeratin immunoprofile differentiates lobular, ductal, and hybrid mammary intraepithelial neoplasias. Hum Pathol. 2002 Jun;33(6):620-7. doi: 10.1053/hupa.2002.124789. PMID 12152161
- [Background] Goldstein NS, Kestin LL, Vicini FA. Clinicopathologic implications of E-cadherin reactivity in patients with lobular carcinoma in situ of the breast. Cancer. 2001 Aug 15;92(4):738-47. PMID 11550142
- [Background] Jacobs TW, Pliss N, Kouria G, Schnitt SJ. Carcinomas in situ of the breast with indeterminate features: role of E-cadherin staining in categorization. Am J Surg Pathol. 2001 Feb;25(2):229-36. doi: 10.1097/00000478-200102000-00011. PMID 11176072
- [Background] Maluf HM, Swanson PE, Koerner FC. Solid low-grade in situ carcinoma of the breast: role of associated lesions and E-cadherin in differential diagnosis. Am J Surg Pathol. 2001 Feb;25(2):237-44. doi: 10.1097/00000478-200102000-00012. PMID 11176073
- [Background] Sullivan ME, Khan SA, Sullu Y, Schiller C, Susnik B. Lobular carcinoma in situ variants in breast cores: potential for misdiagnosis, upgrade rates at surgical excision, and practical implications. Arch Pathol Lab Med. 2010 Jul;134(7):1024-8. doi: 10.5858/2009-0300-OA.1. PMID 20586632
- [Background] Chen YY, Hwang ES, Roy R, DeVries S, Anderson J, Wa C, Fitzgibbons PL, Jacobs TW, MacGrogan G, Peterse H, Vincent-Salomon A, Tokuyasu T, Schnitt SJ, Waldman FM. Genetic and phenotypic characteristics of pleomorphic lobular carcinoma in situ of the breast. Am J Surg Pathol. 2009 Nov;33(11):1683-94. doi: 10.1097/PAS.0b013e3181b18a89. PMID 19701073
- [Background] Bagaria SP, Shamonki J, Kinnaird M, Ray PS, Giuliano AE. The florid subtype of lobular carcinoma in situ: marker or precursor for invasive lobular carcinoma? Ann Surg Oncol. 2011 Jul;18(7):1845-51. doi: 10.1245/s10434-011-1563-0. Epub 2011 Feb 2. PMID 21287281
- [Background] Kuba MG, Murray MP, Coffey K, Calle C, Morrow M, Brogi E. Morphologic subtypes of lobular carcinoma in situ diagnosed on core needle biopsy: clinicopathologic features and findings at follow-up excision. Mod Pathol. 2021 Aug;34(8):1495-1506. doi: 10.1038/s41379-021-00796-9. Epub 2021 Apr 6. PMID 33824462
- [Background] Foschini MP, Miglio R, Fiore R, Baldovini C, Castellano I, Callagy G, Bianchi S, Kaya H, Amendoeira I, Querzoli P, Poli F, Scatena C, Cordoba A, Pietribiasi F, Kovacs A, Faistova H, Cserni G, Quinn C. Pre-operative management of Pleomorphic and florid lobular carcinoma in situ of the breast: Report of a large multi-institutional series and review of the literature. Eur J Surg Oncol. 2019 Dec;45(12):2279-2286. doi: 10.1016/j.ejso.2019.07.011. Epub 2019 Jul 5. PMID 31301938
- See also: Related Info — http://www.cancerscreening.nhs.uk/breastscreen/
- See also: Related Info — http://www.esmo.org